CLINICAL TRIAL: NCT04926740
Title: Balanced Crystalloids (RInger's Lactate) Versus Normal Saline in Adults With Diabetic Ketoacidosis in the Emergency Department: a Pilot Randomized Controlled Trial (BRISK-ED)
Brief Title: Intravenous Fluids in Adults With Diabetic Ketoacidosis in the Emergency Department
Acronym: BRISK-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 119430
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Ketoacidosis
Keywords: randomized controlled trial; emergency department; intravenous fluids; normal saline; Ringer's lactate/balanced crystalloid
MeSH Terms: conditions — Diabetic Ketoacidosis; Emergencies | interventions — Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: This will be a single-centre, triple-blind pilot RCT evaluating the superiority of IV RL (intervention) compared to saline (comparator) in treating adult ED patients presenting with DKA over a one-year period.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patients, treating physicians, and outcome assessors will be blinded to assigned treatment. Our pharmacy will prepare an opaque covering over each fluid bag within study kits, which will not be removed during the infusion to maintain blinding. Each bag will be labelled with a kit number and scannable bar code to ensure the patient receives study fluid as ordered which will be entered on their Medication Administration Record.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ringer's lactate (Experimental): The intervention is administration of IV Ringer's lactate. Rate of study fluid will be at the treating physician's (both ED and inpatient, if consulted for admission) discretion. Apart from fluid administered, there will be no other changes to the patient's clinical care, and patients will receive standard DKA treatment which may include insulin, electrolyte replacement, and/or supportive management. Pharmacy-prepared kits of 8 x 1L bags of study fluid (in Self et al., a maximum of 7090mL was given8) will be kept in a secure space within the ED. Once packaged, IV bags are useable for 30 days before expiration. If a kit is opened but not used completely, individual 1L bags may be returned to the pharmacy to save on costs.
  Interventions: Other: Ringer's lactate
- Normal saline (Active Comparator): The comparator is administration of IV normal saline. Rate of study fluid will be at the treating physician's (both ED and inpatient, if consulted for admission) discretion. Apart from fluid administered, there will be no other changes to the patient's clinical care, and patients will receive standard DKA treatment which may include insulin, electrolyte replacement, and/or supportive management. Pharmacy-prepared kits of 8 x 1L bags of study fluid (in Self et al., a maximum of 7090mL was given8) will be kept in a secure space within the ED. Once packaged, IV bags are useable for 30 days before expiration. If a kit is opened but not used completely, individual 1L bags may be returned to the pharmacy to save on costs.
  Interventions: Other: Ringer's lactate

INTERVENTIONS:
Other: Ringer's lactate — Ringer's lactate is the most commonly used balanced crystalloid. Compared to normal saline, balanced crystalloids have chloride concentrations similar to human plasma; therefore, treatment with balanced crystalloids may lead to faster DKA resolution.
  Other Names: Lactated ringers

SUMMARY:
Diabetes mellitus is a common chronic disease. It is estimated that up to 40% of adults may develop diabetes in their lifetime. Patients with poorly controlled blood sugars often visit the emergency department for treatment of potentially dangerous and life-threatening complications of diabetes, including "diabetic ketoacidosis" (DKA), a condition where the body does not have enough insulin or cannot effectively use the insulin that is produced. As a result, the body produces a chemical called "ketones" as another source of energy, which increase the acid levels of blood and impairs organ function throughout the body.

In the emergency department, patients with DKA are usually treated with insulin and large amounts of intravenous fluid. Recent research suggests the fluid type used may be important in treating DKA. Normal saline (0.9% sodium chloride) is the most commonly used intravenous fluid in treating DKA, but it has a very high concentration of chloride and can lead to additional acid production when given in large volumes. Ringer's lactate is another type of intravenous fluid that more closely matches the chemistry of fluid in our bodies and in theory, does not increase the acidity of blood. While there may be benefits to giving Ringer's lactate instead of normal saline, past studies have included very few patients and thus, definite recommendations on preferred fluid type still cannot be made.

This study's research question is: In adults with DKA, does giving Ringer's Lactate result in faster resolution of DKA compared to normal saline? The investigators hypothesize that patients who are given Ringer's Lactate will have faster resolution of DKA. If the hypothesis is correct, results will provide scientific proof that current diabetic ketoacidosis guidelines should change with respect to fluid choice.

In this study, patients with DKA presenting to the emergency department will be randomly assigned to receive either normal saline or Ringer's Lactate. As this is an exploratory (pilot) study, the main goal is to ensure that a larger study will be practical and feasible on a scale involving multiple emergency departments across Canada. Completion of a larger study across multiple sites with more patients will improve our understanding of how fluid choice influences patient-important outcomes such as faster resolution of DKA (meaning patients can leave hospital sooner), fewer admissions to the intensive care unit, fewer deaths and fewer cases of permanent kidney damage. A total of 52 participants (26 per group) will be recruited for this pilot trial.

This pilot study will assess the practicality of enrolling patients in London and help identify barriers and problems with running a larger trial. The overall goal is to determine if Ringer's Lactate will resolve DKA faster than normal saline. If this is true, patients may spend less time in the hospital, which benefits both individual patients and the healthcare system overall. If this hypothesis is correct, findings could provide high-level proof to change current practice guidelines and affect DKA management globally.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE Diabetic ketoacidosis (DKA) is an acute, life-threatening complication of diabetes which requires treatment with intravenous (IV) fluid and insulin to correct hyperglycemia and reverse acidosis. Current DKA management guidelines recommend normal saline (0.9% sodium chloride) for resuscitation and treatment.1-3 However, saline's chloride content is higher than that of human plasma and can cause a hyperchloremic metabolic acidosis, particularly when administered in large volumes (often needed in patients with DKA). Use of saline may thus worsen the clinical condition of patients who are already in an acidotic state.4-7 Alternatives to saline are balanced crystalloids (e.g. Ringer's lactate-RL) which have chloride concentrations similar to human plasma; therefore, treatment with balanced crystalloids may lead to faster DKA resolution. One recent study (Self et al.) of emergency department (ED) patients presenting with DKA demonstrated that treatment with balanced crystalloids resulted in more rapid DKA resolution compared to saline (13.0 vs 16.9 hours, p=0.004).8 While the difference in resolution time between groups was small, the authors suggested that "consistent implementation of interventions that deliver small improvements in outcomes…can translate into substantial improvements in population health and health system function." However, this study was single-centred, non-blinded, and was a post-hoc subgroup analysis of completed trials (i.e. SMART9 and SALT-ED10) and power was not prospectively calculated. Other studies on this topic have been limited due to small sample sizes (45-77 patients) leading to low power with limited conclusions.11-14

STUDY OBJECTIVE(S); INCLUDING SPECIFIC AIMS AND/OR HYPOTHESES The investigators hypothesize that patients who are administered IV RL will have faster DKA resolution without a concomitant increase in adverse outcomes when compared with normal saline. However, a pilot randomized controlled trial (RCT) is necessary to assess the feasibility of a future multi-centre trial. The specific objectives for this pilot study are to determine the feasibility of conducting a full-scale multi-centred RCT and to use this pilot data to inform the future trial.

METHODS Design and Setting This will be a single-centre, triple-blind pilot RCT evaluating the superiority of IV RL (intervention) compared to saline (comparator) in treating adult ED patients presenting with DKA over a one-year period. The study setting is London Health Sciences Centre (LHSC)'s Victoria Campus, an academic tertiary care centre with ~90,000 ED visits/year in London, Ontario. Study conduct will be in accordance with the CONSORT statement for pilot feasibility trials.15

Study Procedures Screening, Consent, and Enrolment During weekday business hours (M-F 0700-1700), research assistants (RAs) will screen and identify eligible patients using the ED tracking board. They will approach the treating physician to confirm eligibility before discussing the study with the patient and seeking informed consent. Because the diagnosis of DKA requires laboratory confirmation, all patients with a point-of-care blood glucose confirming hyperglycemia (≥14mmol/L) will be approached for enrolment as a "possible DKA patient". If the treating physician agrees that DKA is possible and IV fluid is indicated, study fluid will be administered per the randomization protocol after consent is obtained. If patients are initially enrolled but the physician ultimately confirms they do not meet DKA criteria, they will be excluded from the analysis. During evening and weekend hours, RAs will be available on-call, however nighttime coverage (after 2300h) will not be feasible for this pilot. After hours (and in the event study processes are affected by a prolonged COVID-19 pandemic), treating physicians can directly enroll patients as there will be study posters to outline enrolment processes and physicians will receive email and in-person reminders on study recruitment. Study personnel will review daily ED visit logs to identify missed patients to screen for bias.

Intervention and Comparator The intervention is administration of IV Ringer's lactate and the comparator is administration of IV normal saline. Rate of study fluid will be at the treating physician's (both ED and inpatient, if consulted for admission) discretion. Apart from fluid administered, there will be no other changes to the patient's clinical care, and patients will receive standard DKA treatment which may include insulin, electrolyte replacement, and/or supportive management. Pharmacy-prepared kits of 8 x 1L bags of study fluid (in Self et al., a maximum of 7090mL was given8) will be kept in a secure space within the ED. Once packaged, IV bags are useable for 30 days before expiration. If a kit is opened but not used completely, individual 1L bags may be returned to the pharmacy to save on costs.

Randomization, Blinding, Allocation Concealment Enrolled patients will be block randomized to treatment or comparator in a 1:1 allocation ratio. The block size will be unknown to investigators and those involved in patient care and will be small enough to ensure balance between each arm throughout the trial. The randomization list will be prepared by the pharmacy. The patients, treating physicians, and outcome assessors will be blinded to assigned treatment. The pharmacy will prepare an opaque covering over each fluid bag within study kits, which will not be removed during the infusion to maintain blinding. Each bag will be labelled with a kit number and scannable bar code to ensure the patient receives study fluid as ordered which will be entered on their Medication Administration Record (Figure 1).

DATA COLLECTION Study data for each enrolled patient will be abstracted from the hospital's electronic medical records into the Lawson REDCap data storage platform. Study data will include minimal demographic information (e.g. sex, date of birth), the patient's medical history (e.g. comorbidities, medications), arrival ED information (e.g. CTAS, arrival vitals), hospital interventions (e.g. IV fluids administered), comprehensive bloodwork results, and discharge and outcome information (e.g. length of stay, intubation, diagnosis).

DATA ANALYSIS The investigators will follow an intention-to-treat analysis. Descriptive statistics will be used to summarize patient characteristics. Chi-square tests with 95% confidence intervals will be used to examine differences in categorical variables between groups, and two-tailed unpaired t-tests will be used to compare continuous variables. For this pilot study, no interim analysis, Data Safety Monitoring Board, or adjudication committee is planned, but these will be developed for the full-scale trial. This trial will be registered with ClinicalTrials.gov.

Sample Size The full-scale multi-centred will include 516 participants (258 per arm), assuming α=0.05, power=80%, 1:1 allocation, a 40% (6.76 hours) minimal clinically important reduction in DKA resolution time, and 10% attrition rate. This trial will be conducted at 6 ED sites over 2 years. Based on this, the sample size for this local pilot RCT is 52 participants (26 per arm).

Sample size for Full-Scale Trial The sample size calculation for this trial was based on a study of Clinical Effects of Balanced Crystalloids vs Saline in Adults with Diabetic Ketoacidosis8 which compared the clinical effects of balanced crystalloids with the clinical effects of saline for the acute treatment in DKA in two clinical trials (Isotonic Solutions and Major Adverse Renal Events Trial [SMART]9 and the Saline Against Lactated Ringer's or Plasma-Lyte in the Emergency Department [SALT-ED]10). The primary outcome for this comparison was the time between ED presentation and DKA resolution, measured in hours. Self et al. (2020) found an absolute reduction in time to DKA resolution of 3.9 hours. In the balanced crystalloids group (n=94), the median time to resolution of DKA was 13.0 hrs [IQR: 9.5-18.8], while in the saline group (n=78) the median time to resolution was 16.9 hrs [IQR: 11.9-34.5]. The IQR was used to calculate the standard deviation for each group based on the following assumption for normally distributed data: SD=IQR/1.35. The pooled standard deviation was then calculated based on the sample size and standard deviation of each group from the Self et al. (2020) study [√((n1-1)*SD12 + (n2- 1)*SD22)/(n1+n2-2))] and was determined to be 12.37. To establish superiority of balanced crystalloids versus saline in the time to resolution of DKA, a superiority margin for a clinically significant difference was chosen to be a 40% (=6.76 hours) reduction in time to resolution of DKA based on expert consensus and patient partner feedback. A conservative attrition rate of 10% was selected for the sample size calculation, as loss to follow-up rates should be low given the nature of the intervention (IV fluids) and follow-up period (<24 hours). The actual attrition rate determined by this pilot study will inform the sample size calculation for the full-scale multicentre study. Therefore, to achieve 80% power at the 5% level of significance with equal allocation, the sample size for the balanced crystalloids (Ringer's lactate) group and the saline group, while accounting for a 10% loss to follow up and a 25% reduction in time to DKA resolution, is 516 participants (258 per group). The sample size was calculated using Wang and Ji's (2020) method16 for common clinical study designs available at http://riskcalc.org:3838/samplesize/.

The investigators plan to conduct the full-scale trial at 6 ED sites over 2 years, which would require an average minimum recruitment of 86 participants per site (43 per site per year). This research group has established relationships with these other Canadian EDs and have previously conducted successful studies. If further sites are needed for recruitment, the investigators will leverage the Network of Canadian Emergency Researchers (NCER).

Sample size for Pilot Trial For the full-scale trial, a minimum of 43 participants must be recruited annually per site on average. The LHSC Victoria Campus ED treats approximately 130 patients with DKA annually, based on the hospital's Decision Support data from the most recent fiscal year (Mar 1 2019 - Feb 29 2020).

DKA by Site Patients Victoria Hospital 130 (E1010) Type 1 DM with ketoacidosis 70 (E1110) Type 2 DM with ketoacidosis 51 (E1112) Type 2 DM with keto & lactic acidosis 1 (E1410) Unspecified DM with ketoacidosis 8

Based on research team hours of coverage (0700-2300) and past data from ED presentation time of potentially eligible patients, the investigators expect to approach at least 104 (80%) of eligible patients in the one-year pilot study period, and a minimum of 43 approached participants (41.3%) must be recruited to meet the feasibility target. According to data from similar past trials, the investigators anticipate being able to recruit at least 50% of approached patients (target sample size of 52 patients, 26 in each arm). With 104 patients approached per year, a 90% two-sided confidence interval around the anticipated recruitment rate will have a total width of 0.17, i.e. a lower limit of 0.415 and an upper limit of 0.585. Because the lower limit excludes the minimum feasibility target of 41.3%, the investigators can be 90% confident that the future trial is feasible.

RISKS Participation in this study is entirely voluntary. Patients may refuse to participate, refuse to answer any questions, or withdraw from the study at any time with no effect on their future care. Participants do not waive any legal rights by signing the consent form. They will receive a copy of the letter of information should they be willing to consent.

There are no anticipated risks to participating in this study, other than a low possibility of a privacy breach occurring with the data collected during this study. However, the study team will take all necessary precautions to prevent this from happening and will remove any personal identifiers from all data collection forms.

BENEFITS For participants who are randomized to the Ringer's Lactate Group, there is a possibility that they may benefit from this intervention. The hypothesized benefit from the administration of the IV Ringer's Lactate may include improved faster resolution of DKA than if IV normal saline was administered. However, there is no guarantee that participants will benefit personally from participating in this pilot study.

This study will contribute important knowledge regarding DKA treatment. This pilot study will directly inform if a full-scale clinical trial evaluating the use of a Ringer's Lactate compared to normal saline as part of DKA care in the ED is possible.

ELIGIBILITY:
Inclusion Criteria:

* There are no definitive criteria for diagnosing DKA.3 Thus, using the criteria employed by Self et al.8 and the Diabetes Canada guidelines3 we will include ED patients ≥18 years with a clinical diagnosis and laboratory values consistent with DKA, including:

  * plasma glucose concentration ≥14mmol/L
  * plasma bicarbonate concentration ≤18mmol/L and/or blood pH ≤7.30
  * calculated anion gap >10mmol/L
  * presence of ketones/beta-hydroxybutyrate in serum and/or urine

Exclusion Criteria:

* We will exclude patients who:

  * Are initially seen at another ED and transferred to LHSC for care and/or admission
  * Receive >1L of IV fluid prior to enrolment (e.g. pre-hospital by EMS or while waiting to be seen) - this may cause study contamination
  * Are initially enrolled due to clinical suspicion of DKA based on elevated point-of-care glucose, but ultimately do not meet clinical/laboratory criteria for DKA (e.g. "hyperglycemia" only)
  * Have euglycemic DKA (generally those on SGLT-2 inhibitors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin W Yan, MD, MSc, Principal Investigator — Lawson Health Research Institute/Western University
Locations (1):
- London Health Sciences Centre - Victoria Campus, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitabchi AE, Umpierrez GE, Miles JM, Fisher JN. Hyperglycemic crises in adult patients with diabetes. Diabetes Care. 2009 Jul;32(7):1335-43. doi: 10.2337/dc09-9032. No abstract available. PMID 19564476
- [Background] Roberts A, James J, Dhatariya K; Joint British Diabetes Societies (JBDS) for Inpatient Care. Management of hyperglycaemia and steroid (glucocorticoid) therapy: a guideline from the Joint British Diabetes Societies (JBDS) for Inpatient Care group. Diabet Med. 2018 Aug;35(8):1011-1017. doi: 10.1111/dme.13675. PMID 30152586
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Goguen J, Gilbert J. Hyperglycemic Emergencies in Adults. Can J Diabetes. 2018 Apr;42 Suppl 1:S109-S114. doi: 10.1016/j.jcjd.2017.10.013. No abstract available. PMID 29650082
- [Background] Myburgh JA, Mythen MG. Resuscitation fluids. N Engl J Med. 2013 Sep 26;369(13):1243-51. doi: 10.1056/NEJMra1208627. No abstract available. PMID 24066745
- [Background] Casey JD, Brown RM, Semler MW. Resuscitation fluids. Curr Opin Crit Care. 2018 Dec;24(6):512-518. doi: 10.1097/MCC.0000000000000551. PMID 30247219
- [Background] Morgan TJ, Venkatesh B, Hall J. Crystalloid strong ion difference determines metabolic acid-base change during acute normovolaemic haemodilution. Intensive Care Med. 2004 Jul;30(7):1432-7. doi: 10.1007/s00134-004-2176-x. Epub 2004 Feb 28. PMID 14991093
- [Background] Omron EM, Omron RM. A physicochemical model of crystalloid infusion on acid-base status. J Intensive Care Med. 2010 Sep;25(5):271-80. doi: 10.1177/0885066610371633. PMID 20622258
- [Background] Self WH, Evans CS, Jenkins CA, Brown RM, Casey JD, Collins SP, Coston TD, Felbinger M, Flemmons LN, Hellervik SM, Lindsell CJ, Liu D, McCoin NS, Niswender KD, Slovis CM, Stollings JL, Wang L, Rice TW, Semler MW; Pragmatic Critical Care Research Group. Clinical Effects of Balanced Crystalloids vs Saline in Adults With Diabetic Ketoacidosis: A Subgroup Analysis of Cluster Randomized Clinical Trials. JAMA Netw Open. 2020 Nov 2;3(11):e2024596. doi: 10.1001/jamanetworkopen.2020.24596. PMID 33196806
- [Background] Semler MW, Self WH, Wanderer JP, Ehrenfeld JM, Wang L, Byrne DW, Stollings JL, Kumar AB, Hughes CG, Hernandez A, Guillamondegui OD, May AK, Weavind L, Casey JD, Siew ED, Shaw AD, Bernard GR, Rice TW; SMART Investigators and the Pragmatic Critical Care Research Group. Balanced Crystalloids versus Saline in Critically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):829-839. doi: 10.1056/NEJMoa1711584. Epub 2018 Feb 27. PMID 29485925
- [Background] Self WH, Semler MW, Wanderer JP, Wang L, Byrne DW, Collins SP, Slovis CM, Lindsell CJ, Ehrenfeld JM, Siew ED, Shaw AD, Bernard GR, Rice TW; SALT-ED Investigators. Balanced Crystalloids versus Saline in Noncritically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):819-828. doi: 10.1056/NEJMoa1711586. Epub 2018 Feb 27. PMID 29485926
- [Background] Mahler SA, Conrad SA, Wang H, Arnold TC. Resuscitation with balanced electrolyte solution prevents hyperchloremic metabolic acidosis in patients with diabetic ketoacidosis. Am J Emerg Med. 2011 Jul;29(6):670-4. doi: 10.1016/j.ajem.2010.02.004. Epub 2010 May 1. PMID 20825879
- [Background] Van Zyl DG, Rheeder P, Delport E. Fluid management in diabetic-acidosis--Ringer's lactate versus normal saline: a randomized controlled trial. QJM. 2012 Apr;105(4):337-43. doi: 10.1093/qjmed/hcr226. Epub 2011 Nov 22. PMID 22109683
- [Background] Yung M, Letton G, Keeley S. Controlled trial of Hartmann's solution versus 0.9% saline for diabetic ketoacidosis. J Paediatr Child Health. 2017 Jan;53(1):12-17. doi: 10.1111/jpc.13436. PMID 28070957
- [Background] Williams V, Jayashree M, Nallasamy K, Dayal D, Rawat A. 0.9% saline versus Plasma-Lyte as initial fluid in children with diabetic ketoacidosis (SPinK trial): a double-blind randomized controlled trial. Crit Care. 2020 Jan 2;24(1):1. doi: 10.1186/s13054-019-2683-3. PMID 31898531
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Wang X, Ji X. Sample Size Estimation in Clinical Research: From Randomized Controlled Trials to Observational Studies. Chest. 2020 Jul;158(1S):S12-S20. doi: 10.1016/j.chest.2020.03.010. PMID 32658647
- [Derived] Yan JW, Slim A, Van Aarsen K, Choi YH, Byrne C, Poonai N, Collins H, Clemens KK. Balanced crystalloids (RInger's lactate) versus normal Saline in adults with diabetic Ketoacidosis in the Emergency Department (BRISK-ED): a pilot randomised controlled trial. Emerg Med J. 2024 Jan 22;41(2):103-111. doi: 10.1136/emermed-2023-213290. PMID 38050056
- [Derived] Yan JW, Slim A, Van Aarsen K, Choi YH, Byrne C, Poonai N, Collins H, Clemens KK. Balanced crystalloids (RInger's lactate) versus normal Saline in adults with diabetic Ketoacidosis in the Emergency Department (BRISK-ED): a protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2023 Jul 13;9(1):121. doi: 10.1186/s40814-023-01356-5. PMID 37443083

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We approached 74 patients for consent during the study period at our site and 8 declined participation.
Period: Overall Study
Arm/Group | Ringer's Lactate | Normal Saline
Started | 34 | 32
Completed | 25 | 27
Not Completed | 9 | 5
Not completed — Ineligible: received >1L of pre-study fluid prior to enrolment | 2 | 1
Not completed — Ineligible: subsequently found to not have true DKA | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ringer's Lactate | Normal Saline | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [33 to 65] | 43 [24 to 59] | 46 [25 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 16 | 15 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diabetes type [Count of Participants; unit: Participants]
  Type 1 | 9 | 17 | 26
  Type 2 | 14 | 8 | 22
  New diagnosis | 2 | 2 | 4
Comorbidities [Number; unit: participants]
  Psychiatric illness | 10 | 11 | 21
  Hypertension | 9 | 12 | 21
  Dyslipidemia | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Patient Recruitment Rate (Feasibility Outcome)
Description: The primary feasibility outcome is patient recruitment rate over the one-year study period. We will also measure adherence to the protocol for this pilot study. This pilot is not powered to determine differences in treatment groups; however, a priori outcome definition and accurate outcome assessment is needed to inform the future study.
Time Frame: One year
Population: We approached 74 patients for consent and 8 declined participation. Ultimately, we randomized 66 patients to receive RL (34 patients) or NS (32 patients); thus, our recruitment rate was 66/74 (89.2%).
Measure: Count of Participants; unit: Participants
Groups:
- Patient Recruitment Rate: Feasibility outcome
Arm/Group | Patient Recruitment Rate
Number analyzed (Participants) | 74
Participants | 66

2. Primary Outcome: Time to DKA Resolution (Efficacy Outcome)
Description: Time to DKA resolution (hours), defined as the time elapsed between ED presentation and ketoacidosis resolution, following criteria from the American Diabetes Association Consensus Statement on Hyperglycemic Crises1 (plasma glucose <11.1 mmol/L and two of: plasma bicarbonate ≥15mmol/L, venous pH >7.3 or anion gap ≤12mmol/L).
Time Frame: Up to 48 hours
Population: Of 66 overall patients consented, 14 were subsequently excluded upon further review as they did not meet criteria for DKA or received greater than 1 litre of fluid before randomization, leaving 52 included patients in our study. Due to a pharmacy error with respect to the allocation list for one patient, there were 25 patients in the RL group and 27 in the NS group.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Normal Saline | Ringer's Lactate
Number analyzed (Participants) | 27 | 25
hours | 12.7 [7.9 to 19.2] | 15.7 [10.4 to 18.8]

3. Secondary Outcome: Time to Insulin Infusion Discontinuation
Description: Time to insulin infusion discontinuation
Time Frame: Up to 48 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Ringer's Lactate | Normal Saline
Number analyzed (Participants) | 25 | 27
hours | 15.9 [5.7 to 39.2] | 15.5 [6.7 to 36.4]

4. Secondary Outcome: Intensive Care Unit Admission
Description: Intensive care unit admission
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ringer's Lactate | Normal Saline
Number analyzed (Participants) | 25 | 27
Participants | 1 | 1

5. Secondary Outcome: In-hospital Death
Description: In-hospital death
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ringer's Lactate | Normal Saline
Number analyzed (Participants) | 25 | 27
Participants | 0 | 0

6. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Ringer's Lactate | Normal Saline
Number analyzed (Participants) | 25 | 27
hours | 3.3 [2.0 to 6.1] | 1.4 [0.3 to 5.8]

7. Secondary Outcome: Hyper- or Hypo-kalemia Post-emergency Department
Description: >6.0 or <3.0 mmol/L
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ringer's Lactate | Normal Saline
Number analyzed (Participants) | 25 | 27
Participants | 24 | 12

8. Secondary Outcome: In-hospital Acute Kidney Injury (Stage 2 or Greater) Post-emergency Department
Description: Serum creatinine increase >200% from baseline or <0.5mL/kg/hr urine output for <12 hours
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ringer's Lactate | Normal Saline
Number analyzed (Participants) | 25 | 27
Participants | 4 | 3

9. Secondary Outcome: Major Adverse Kidney Events
Description: Composite of i) death, ii) new renal replacement therapy, iii) final serum creatinine >/= 200% baseline at the earliest of hospital discharge or 30 days after ED presentation
Time Frame: 30 days
Measure: Number; unit: events
Arm/Group | Ringer's Lactate | Normal Saline
Number analyzed (Participants) | 25 | 27
events | 4 | 2

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse event = death, intensive care unit admission, intubation, in-hospital acute kidney injury, and major adverse kidney events at 30 days
Arm/Group | Ringer's Lactate | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 7/25 | 4/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ringer's Lactate (N=25) | Normal Saline (N=27)
Major adverse kidney event within 30 days of ED presentation (Renal and urinary disorders) | 4 (4) | 2 (2)
Intensive Care Unit Admission (General disorders) | 1 (1) | 1 (1)
Intubation (Surgical and medical procedures) | 2 (2) | 0 (0)
Acute kidney injury (in-hospital) (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT04926740/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT04926740/ICF_001.pdf